CLINICAL TRIAL: NCT00212368
Title: Phase3,Open-label,Clinical Trial of Zinc Acetate for Treatment of Wilson's Disease in Japan.
Brief Title: Efficacy and Safety Study of Zinc Acetate to Treat Wilson's Disease in Japan.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nobelpharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-02-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Wison's Disease
MeSH Terms: interventions — Zinc Acetate

INTERVENTIONS:
Drug: Zinc acetate

SUMMARY:
The purpose of this study is to determine whether Zinc Acetate is effective and safe in the treatment of Wilson's disease among Japanese.

ELIGIBILITY:
Inclusion Criteria:

* Wilson's disease(adult,infant,pregnant woman)

Exclusion Criteria:

* acute hepatitis
* malignant tumor

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-10; Primary Completion 2005-08 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koudou Ishii, M.D., Study Director — National MINAMIYOKOHAMA Hospital